CLINICAL TRIAL: NCT05818098
Title: A Prospective, Multicenter Clinical Trial in Evaluating the Safety and Efficacy of the Intravascular Lithotripsy System in Patients With Coronary Artery Calcification
Brief Title: Coronary Intravascular Lithotripsy System in Patients With Coronary Artery Calcification (VIGOUR)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai MicroPort Rhythm MedTech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AMD-D-002
Record Dates: First submitted 2023-04-05; First posted 2023-04-18 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2022-11

CONDITIONS: Coronary Artery Calcification
Keywords: calcification; coronary artery
MeSH Terms: conditions — Calcinosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intravascular Lithotripsy System (Experimental): Subjects in experimental group will be treated with the Intravascular Lithotripsy System manufactured by Shanghai Microport Rhythm Co. Ltd.
  Interventions: Device: Intravascular Lithotripsy System of Shanghai MicroPort Rhythm

INTERVENTIONS:
Device: Intravascular Lithotripsy System of Shanghai MicroPort Rhythm — The Intravascular Lithotripsy System is a single-use, sterile, disposable balloon angioplasty catheter that contains a series of unfocused, electrohydraulic lithotripsy emitters, which convert electrical energy into transient acoustic circumferential pressure pulses that disrupt both superficial and deep calcium within vascular plaque.

SUMMARY:
This is a prospective and multicenter clinical investigation aiming to evaluate the safety and effectiveness of coronary intravascular lithotripsy system for the treatment of patients with coronary calcification.

DETAILED DESCRIPTION:
This trial is a prospective and multicenter clinical trial. 189 subjects are expected to be recruited in 20 research centers in China.

1. All subjects with coronary calcified lesions participating in this clinical study must have only one lesion length of no more than 40 mm and located in an coronary artery with a diameter of ≥ 2.00 mm but ≤ 4.00 mm.
2. All subjects receive clinical follow-up during hospitalization, 30 days and 6 months after surgery.

ELIGIBILITY:
Inclusion Criteria:

Clinical Inclusion Criteria:

1. Subjects aged between 18 and 85.
2. Subjects who can undergo percutaneous coronary intervention (PCI).
3. Subjects with asymptomatic evidence of ischemia, stable or unstable angina pectoris, or old myocardial infarction.
4. Left Ventricular Ejection Fraction (LVEF) ≥30% as measured by echocardiography for subjects within 6 months before enrollment. (In case of multiple LVEF results, the data closest to the baseline procedure was taken.)
5. Subjects who are able to understand the purpose of the trial, participate voluntarily or by proxy and indicate by signing the informed consent form that they recognize the risks and benefits described in the informed consent document and are willing to undergo clinical follow-up.

Angiography Inclusion Criteria:

1. There is only one target lesion that needs to be treated.
2. The target lesion must be located in a de novo native coronary artery with a reference vessel diameter (RVD) ≥2.00 mm to ≤4.00 mm as visually measured.
3. The target lesion angiography shows a stenosis rate ranging from ≥70% (visually measured) or ≥50% to <70% with symptoms of ischemia.

   Ischemic symptoms were defined as any of the following:
   * Exercise stress test positive
   * Fractional Flow Reserve (FFR) ≤ 0.8 or iFR < 0.9
   * Minimum lumen area (MLA) ≤ 4.0 mm2 by IVUS or OCT
4. The target lesion length must be less than 40 mm (visually measured).
5. The target lesion must meet one of the following :

   * During angiography, clear hyperdense opacities can be observed on both sides of the arterial wall when the heart pulsates and does not pulsate
   * Presence of calcium of ≥270°at one cross-section via IVUS or OCT
6. Target lesion TIMI flow 3 prior to the use of the test device (at baseline or after balloon pre-dilatation).
7. The lesion that 0.014 "guidewire can cross.

Exclusion Criteria:

General Exclusion Criteria:

1. Subjects who present with AMI recently (within 7 days)
2. Subjects who have hemodynamic instability or a severe reduction in activity tolerance (NYHA cardiac function Grade Ⅲ, Ⅳ).
3. Subjects who have an intra-cardiac thrombus as shown by echocardiography within 30 days before enrollment.
4. Subjects who have already received or are waiting for organ transplantation.
5. Subjects who are receiving or scheduled to receive chemotherapy within 30 days before or after the baseline procedure.
6. Subjects who have a platelet count < 60 x 10^9/L or > 750 x 10^9/L or other hemorrhagic diathesis, coagulation dysfunction, blood transfusion resistance.
7. Subjects who have severe hepatic dysfunction (transaminases more than 3 times the upper limit of normal).
8. Subjects who have chronic renal failure and a serum creatinine level > 2.5 mg/Dl (or 221µmol/L).
9. Subjects who have active peptic ulcer diseases or active gastrointestinal (GI) bleeding within 6 months before enrollment.
10. Subjects who are unable to receive dual antiplatelet therapy for at least 6 months due to various reasons.
11. Subjects who experience cerebrovascular accident (CVA) or transient ischemic attack (TIA) within the past six months, or have permanent neurological defects that may cause nonconformity with the protocol.
12. Subjects who plan to undergo rotational atherectomy, cutting balloon, scored balloon, or laser coronary atherectomy during the baseline procedure.
13. Subjects who have received stent placement for target vessel (including collateral branches) within 12 months prior to the baseline procedure.
14. Subjects who have received any type of PCI treatment for non-target vessels within 24 hours prior to the baseline procedure.
15. Subjects who are scheduled to receive a cardiac intervention or cardiac surgery within 30 days of the index procedure.
16. Subjects who have been treated with intracoronary brachytherapy at any time previously.
17. Subjects who are allergic to investigational stent system or concomitant drugs required in the protocol (such as everolimus, sirolimus, or structure-related compounds; fluorine-containing polymers; antiplatelet agents such as aspirin, ticagrelor, or thienopyridines; contrast agent; narcotics).
18. Subjects with other serious medical conditions (such as cancer) may shorten their life expectancy to less than 12 months.
19. Subjects who plan to undergo a procedure that may lead to non-conformity with the protocol or confusion in data interpretation.
20. Subjects who are participating in another investigational drug or device clinical trial in which the primary endpoint is still not reached, or intend to participate in another investigational drug or device clinical trial within 6 months after baseline procedure.
21. Pregnant or breast-feeding subjects (women who may become pregnant must receive a pregnancy test within seven days prior to the baseline procedure).
22. Subjects who are found to have poor compliance and unable to complete the trial as required as judged by the investigators.

Angiography Exclusion Criteria:

1. Subjects with target lesions meet the following criteria:

   * Target lesions located within or involving 5 mm of the ostium of the left and right main coronary arteries (LAD/LCX/RCA);
   * Target lesions that involve bifurcation lesions (bifurcation lesion ostial diameter stenosis greater than 30%);
   * Entering through a great saphenous vein graft or an artery graft;
   * Target lesions with thrombosis or suspected thrombosis;
   * Target vessel with C-F type dissection according to NHLBI classification following pre-procedure angiography or guidewire crossing;
   * In-stent restenosis involved in target lesions.
2. Subjects with unprotected left main coronary artery diseases (diameter stenosis >30%).
3. Subjects with other clinically significant lesions at target vessels (diameter stenosis >50%).
4. The target vessel (including collateral) near the target lesion or within 10 mm (visually) from the distal end of the target lesion has received stent implantation at any time before baseline surgery.
5. Subjects with lesions that guide wire cannot pass through or retrieve due to various reasons (such as serious distortion at the proximal target vessel).

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 189 (Estimated)
Dates: Start 2023-03-29 (Actual); Primary Completion 2023-09 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Procedure success | During hospitalization (up to 7 days after procedure)
  Procedure success is defined as the ability of intravascular lithotripsy (IVL) to produce residual diameter stenosis ≤30% after stenting with no evidence of in-hospital MACE (maximum of 7 days) (MACE: defined as the composite of cardiac death, myocardial infarction, and target vessel revascularization)

SECONDARY OUTCOMES:
Device success | Baseline procedure
  Device success is defined as delivery of the IVL catheter across the target lesion and delivery of lithotripsy without serious angiographic complications immediately after IVL.
Angiographic success | Baseline procedure
  Angiographic success is defined as stent delivery with ≤30% residual stenosis and without serious angiographic complications.
MACE freedom rate at 30 days after the index procedure | within 30 days of baseline procedure
  MACE is defined as a composite of cardiac death, myocardial infarction[MI], and target vessel revascularization [TVR].
  (Periprocedural MI is defined as peak post-PCI CK-MB level >3 x the upper limit of normal [ULN], both non-Q wave myocardial infarction or Q-wave myocardial infarction.)
Procedure-related serious complications | Baseline procedure
  Procedure-related serious complications included severe dissection (Type D-F, according to NHLBI classification system), perforation, abrupt closure, and persistent slow flow/no-reflow during the baseline procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Bo Yu, M.D., Principal Investigator — The Second Affiliated Hospital of Harbin Medical University
Locations (1):
- The Second Affliated Hospital Ha'erbin Medical University, Harbin, Heilongjiang, China